CLINICAL TRIAL: NCT01321424
Title: Investigator Sponsored, Pilot Study to Assess the Diurnal Variation in Tear Osmolarity as a Predictor of Dry Eye Disease Etiology
Brief Title: Diurnal Variation in Tear Osmolarity
Status: Completed | Type: Observational
Sponsor: Ophthalmic Consultants of Long Island (Other)
Collaborators: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: ALRGN01
Record Dates: First submitted 2011-03-21; First posted 2011-03-23 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: Dry Eye Disease
Keywords: Dry Eye; Tear Osmolarity; Meibomain Gland Disease; Aqueous Dificiency; Tear film abnormality
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Aqueous Dificiency Dry Eye: 20 Participants
- Meibomian Gland Disease Dry Eye: 20 Participants
- Normal Eye: 20 Participants

SUMMARY:
The purpose of this study is to measure the change in Tear Osmolarity during the course of the day to support clinical diagnosis of aqueous deficiency or meibomian gland disease and differentiate between the two forms of dry eye.

DETAILED DESCRIPTION:
The premise of this study is that dry eye disease, specifically tear osmolarity, changes during the course of the day based on the etiology of the dry eye and that aqueous-deficiency dry eye will worsen during the course of the day while meibomian gland deficiency will stabilize or possibly even improve during the course of the day.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and females ≥ 18 years old
2. Negative urine pregnancy results for females of childbearing potential
3. Able to read and sign an informed consent form and show willingness to comply with the study protocol visits and procedures
4. Has 20/40 BCVA or better in at least one eye
5. Does not currently wear contact lenses
6. For Aqueous-Deficiency Group:

   * Has symptoms of Dry Eye
   * Schirmer testing ≤ 10 mm
   * Tear Break Up Time ≤ 8 seconds
   * Conjunctival staining ≥ 1+
   * Meibomian gland inspissations ≤ 1+
   * No lid thickening, lid erythema, or thickened, turbid meibomian gland secretions
7. For Meibomian Gland Disease Group:

   * Has symptoms of Dry Eye
   * Schirmer testing ≥ 10 mm
   * Tear Break Up Time ≤ 8 seconds
   * Conjunctival staining ≥ 1+
   * Meibomian gland inspissations ≥ 2+
8. For Normal Group:

   * Has no symptoms of Dry Eye
   * Schirmer testing > 10 mm
   * Tear Break Up Time > 8 seconds
   * No or trace Conjunctival staining
   * No Meibomian gland inspissations

Exclusion Criteria:

1. Any topical medication within the last three months, except for artificial tears
2. Unable to discontinue use of artificial tears during the course of the day for Visit 2
3. Any Systemic disease, which in the opinion of the Investigator, may affect ocular health or confound study results
4. Any active ocular disease other than Dry Eye Disease, Meibomian Gland Disease or Sjogren's Syndrome, which in the opinion of the Investigator, may affect ocular health or confound study results
5. Clinically significant lid or conjunctival abnormalities, neovascularization, corneal scars or corneal opacities
6. Clinically significant limbal or bulbar injection, or corneal staining not due to DES
7. Has worn hard or rigid gas permeable contact lenses within 1 year
8. Has worn soft contact lenses within 1 week
9. Has had eye surgery or an eye injury within 6 months
10. Positive urine pregnancy results for females of childbearing potential
11. Any changes in current medication within 30 days of Visit 2 or anticipated change during course of study, which in the opinion of the Investigator may confound study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care facility
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-03; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
The measured difference in Tear Osmolarity during the course of the day to support clinical diagnosis and differentiate between aqueous-deficiency and meibomian gland disease. | 1 Day (AM and PM Diurnal)

SECONDARY OUTCOMES:
Ocular Improvement | 31 Days
  Improvement in Ocular Surface Disease Index, Best Corrected Visual Acuity, Uncorrected Visual Acuity, Slit Lamp Exam, Schirmer test, Lissamine green conjunctival staining, Fluorescein corneal staining and Tear Break Up Time

CONTACTS AND LOCATIONS:
Overall Officials: Eric D Donnenfeld, MD, Principal Investigator — Ophthalmic Consultants of Long Island; Barbara Burger, RN, Study Director — Ophthalmic Consultants of Long Island
Locations (6):
- United States (6):
  - Ophthalmic Consultants of Connecticut, Fairfield, Connecticut
  - Ophthalmic Consultants of Long Island, Lynbrook, New York
  - Ophthalmic Consultants of Long Island, Manhasset, New York
  - Ophthalmic Consultants of Long Island, Port Jefferson, New York
  - Ophthalmic Consultants of Long Island, Rockville Centre, New York
  - Ophthalmic Consultants of Long Island, Valley Stream, New York

IPD SHARING:
Plan to Share IPD: Yes
PI will present study outcomes to associates